CLINICAL TRIAL: NCT01458561
Title: An Investigational Plan Evaluating the Operative Management of Parenchymal Bleeding By Means of an Adjunctive Application of BioFoam Surgical Matrix in Liver Surgery
Brief Title: Adjunctive Application of BioFoam Surgical Matrix in Liver Surgery
Acronym: BARRIER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor terminated due to signif. difficulty with pilot investigation enrollment
Sponsor: CryoLife, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: CryoLife (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BFM0801-C
Record Dates: First submitted 2011-06-07; First posted 2011-10-25 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Intraoperative Bleeding
Keywords: Hemostatic agent; Liver surgery; Hemostasis
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BioFoam Surgical Matrix (Experimental): Control of bleeding using BioFoam Surgical Matrix as a surgical adjunct
  Interventions: Device: BioFoam Surgical Matrix
- Gelfoam Plus (Active Comparator): Control of bleeding using Gelfoam Plus as a surgical adjunct
  Interventions: Device: Gelfoam Plus

INTERVENTIONS:
Device: BioFoam Surgical Matrix — Surgical adjunct to control bleeding in open liver surgery
  Other Names: BioFoam
  Arms: BioFoam Surgical Matrix
Device: Gelfoam Plus — Surgical adjunct in control of bleeding in open liver surgery
  Other Names: Gelfoam with thrombin
  Arms: Gelfoam Plus

SUMMARY:
This is a prospective, multicenter, randomized, controlled investigation. Subjects in which bleeding from the exposed parenchymal surface is observed intraoperatively following the ligature of vessels visible with the unaided eye will be randomized to an adjunctive application of BioFoam or a standard topical hemostatic agent (Gelfoam with thrombin, in the form of Gelfoam Plus) to the entire exposed parenchymal surface. Following primary treatment of the exposed parenchymal surface as prescribed by the randomization scheme, treatment sites will be visually evaluated for the continued presence of bleeding. The overall objective of this investigation is to collect clinical data concerning the safety and effectiveness of BioFoam used as an adjunct to conservative measures of achieving hemostasis, such as manual pressure, cautery, and ligation, for intraoperative capillary, arteriolar, and venular bleeding (5 second stack of 5 gauze surface "Bleeding Score" = 1b or 2, score to be validated) on newly resected liver parenchyma in hemodynamically stable (American College of Surgeons' Advanced Trauma Life Support Class I Hemorrhage) and non-coagulopathic patients in the open treatment of exposed liver parenchyma versus a standard topical hemostatic agent, Gelfoam Plus. It is not intended for traumatic liver injury. The investigation will be conducted at a maximum of three investigational sites.

ELIGIBILITY:
Preoperative Inclusion Criteria:

* Subject is undergoing an elective liver resection procedure that requires treatment of the exposed parenchymal surface due to the intraoperative presence of blood following ligature of vessels visible with the unaided eye;
* Subject has adequate hepatic function as indicated by a Model for End-Stage Liver Disease (MELD) score of <10 at ≤30 days and at ≤7 days prior to surgery;
* Subject has adequate hemostatic function identified as an international normalized ratio (INR), platelet count, and activated clotting time within the central laboratory's normal reference range;
* Subject or an authorized legal representative is willing and able to give prior written informed consent for investigation participation; and
* Subject is ≥ 18 years of age.

Preoperative Exclusion Criteria:

* Subject with known or suspected sensitivity to products of bovine origin
* Subject with known or suspected sensitivity to glutaraldehyde
* Subject with active infection (either systemic or in the treatment region) or hepatic cysts due to parasitic disease and/or abscesses due to bacterial and/or amebic disease;
* Subject with abnormal calcium metabolism identified as values for ionized calcium and serum calcium corrected for serum albumin that are outside of the central laboratory's normal reference range;
* Subject with abnormal renal status identified as an estimated glomerular filtration rate (eGFR), blood urea nitrogen (BUN), serum creatinine, sodium, chloride, potassium, and/or bicarbonate values that are outside of the central laboratory's normal reference range;
* Subject with hyperparathyroidism identified as an intact parathyroid hormone level >72 pg/mL, serum calcium >10.6 mg/dL, and phosphate <2.4 mg/dL, and, for secondary or tertiary hyperparathyroidism only, alkaline phosphatase >147 U/L
* Subject with a pancreatic amylase and/or lipase value outside of the central laboratory's normal reference range;
* Subject with blunt and/or penetrating liver trauma;
* Subject diagnosed with any coagulation disorder;
* Subject whose life-expectancy is less than that required for the prescribed follow-up duration;
* Subject who has been treated with an investigational product and has not completed the entire follow-up period for that investigational product;
* Subject with any surgical implant that would interfere with necessary follow-up imaging;
* Subject who is pregnant (as confirmed by a urine pregnancy test), planning on becoming pregnant during the follow-up period, or actively breast-feeding;
* Subject who is undergoing concomitant procedures other than (1) cholecystectomy, (2) umbilical hernia repair, or (3) uncomplicated colon resection (i.e., no significant spillage);
* Subject who is immunocompromised;
* Subject with an American Society of Anesthesiologist (ASA) Score >2
* Subject with a MELD score of ≥10 at ≤30 days or at ≤7 days prior to surgery;
* Subject diagnosed with an autoimmune disease; and
* Subject in whom the surgeon intends to use adhesion prevention products.
* Subject who is returning to the operating room (OR) to address a complication associated with a liver resection, including but not limited to hematoma evacuation and biliary leak.

Intraoperative Inclusion Criterion:

- Subject in whom bleeding (assignment of a "Bleeding Score" of 1 or 2) from the exposed parenchymal surface after ligature of vessels visible with the unaided eye and removal of any clamps used for hemostasis is observed

Intraoperative Exclusion Criterion:

- Subject in whom any major intraoperative bleeding incidences during the resection procedure occurred (i.e., subject with assignment of an American College of Surgeons Advanced Trauma Life Support Hemorrhage Class of II, III, or IV Hemorrhage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Capps, MS, Study Director — CryoLife, Inc.
Locations (2):
- United States (2):
  - Stanford University Medical Center, Palo Alto, California
  - Swedish Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was limited to potential subjects who were being seen by a liver surgeon because they required a liver resection procedure. The first site was cleared to begin recruitment on October 20, 2010 and recruitment was closed on August 31, 2012 when all investigators were formally notified of the decision to terminate the study.
Pre-assignment Details: All potential subjects were required to meet preoperative and operative screening criteria in order to be enrolled into the investigation and assigned to a treatment group.
Groups:
- BioFoam Surgical Matrix: Control of bleeding using BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Gelfoam Plus: Control of bleeding using Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Period: Overall Study
Arm/Group | BioFoam Surgical Matrix | Gelfoam Plus
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BioFoam Surgical Matrix | Gelfoam Plus | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 57 (0) | 57 (0)
Gender [Number; unit: participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Intraoperative Hemostasis Following Open Liver Resection Surgery in Subjects Receiving an Application of BioFoam or a Standard Topical Hemostatic Agent
Description: Number of subjects achieving intraoperative hemostasis (y/n) at 3 minutes following a single application of the prescribed hemostatic agent
Time Frame: 3 minutes following a single application of the prescribed hemostatic agent
Population: Study was terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: participants
Groups:
- Control Bleeding in BioFoam Subjects/Participants: Control of bleeding in subjects/participants who receive BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Control Bleeding in Gelfoam Plus Subjects/Participants: Control of bleeding in subjects/participants who receive Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Control Bleeding in BioFoam Subjects/Participants | Control Bleeding in Gelfoam Plus Subjects/Participants
Number analyzed (Participants) | 0 | 1
participants |  | 1

2. Secondary Outcome: Time to Hemostasis
Description: Number of subjects achieving hemostasis [by assessing for hemostasis (yes/no)] at pre-determined time points: 1, 3, 5, 7, and 10 minutes following application of prescribed hemostatic agent. Time to hemostasis is recorded as the first of the predetermined time points to receive a "yes" assessment.
Time Frame: 1, 3, 5, 7, and 10 minutes following application of prescribed hemostatic agent
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: minutes
Groups:
- Subjects/Participants Receiving BioFoam: Number of subjects achieving hemostasis (y/n) at predetermined time points (1, 3, 5, 7, 10 min) in subjects/participants receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Subjects/Participants Receiving Gelfoam Plus: Number of subjects achieving hemostasis (y/n) at predetermined time points (1, 3, 5, 7, 10 min) in subjects/participants receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Subjects/Participants Receiving BioFoam | Subjects/Participants Receiving Gelfoam Plus
Number analyzed (Participants) | 0 | 1
minutes |  | 1

3. Secondary Outcome: Achievement of Immediate Hemostasis
Description: Number of subjects achieving hemostasis at 1 minute after application of prescribed hemostatic agent
Time Frame: 1 minute after application of prescribed hemostatic agent
Population: Study was terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: participants
Groups:
- Achieve Immediate Hemostasis in BioFoam Subjects/Participants: Number of subjects achieving immediate hemostasis (1 minute following application of hemostatic agent) in subjects/participants receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Achievement of Immediate Hemostasis in Gelfoam Plus Subjects: Number of subjects achieving immediate hemostasis (1 minute following application of hemostatic agent) in subjects/participants receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Achieve Immediate Hemostasis in BioFoam Subjects/Participants | Achievement of Immediate Hemostasis in Gelfoam Plus Subjects
Number analyzed (Participants) | 0 | 1
participants |  | 1

4. Secondary Outcome: Intraoperative Blood Loss
Description: Amount of blood lost between time of initial application of prescribed hemostatic agent and confirmed achievement of hemostasis (achievement of hemostasis eval. out to 10 minutes following application of prescribed hemostatic agent)
Time Frame: Time from initial application to confirmed achievement of hemostasis (eval. up to 10 minutes following application of hemostatic agent)
Population: Study terminated before appropriate data collection/analysis
Groups:
- Intraop. Blood Loss in BioFoam Surgical Matrix Subjects: Amount of blood lost intraoperatively in subjects receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Intraop. Blood Loss in Gelfoam Plus Subjects: Amount of blood lost intraoperatively in subjects receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Intraop. Blood Loss in BioFoam Surgical Matrix Subjects | Intraop. Blood Loss in Gelfoam Plus Subjects
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Amount of Postoperative Bilious Drainage
Time Frame: Time from drain insertion to drain removal (where applicable), average 24-72 hours postoperatively
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: milliliters (mL)
Arm/Group | BioFoam Surgical Matrix | Gelfoam Plus
Number analyzed (Participants) | 0 | 1
milliliters (mL) |  | NA — Study terminated before appropriate data collection/analysis

6. Secondary Outcome: Amount of Postoperative Fluid Loss
Description: Amount of fluid lost postoperatively [measured between time of drain insertion (if applicable) to drain removal, average 24-72 hours postoperatively]
Time Frame: Time from drain insertion to drain removal (where applicable), average 24-72 hours postoperatively
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: milliliters (mL)
Arm/Group | BioFoam Surgical Matrix | Gelfoam Plus
Number analyzed (Participants) | 0 | 1
milliliters (mL) |  | NA — Study terminated before appropriate data collection/analysis

7. Secondary Outcome: Duration of Drainage
Description: Total length of time between drain insertion and last recorded emptying time during hospitalization (where applicable), average 24-72 hours postoperatively
Time Frame: Time between drain insertion and last recorded emptying time during hospitalization (where applicable), average 24-72 hours postoperatively
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: hours
Groups:
- Duration of Postoperative Drainage in BioFoam Subjects: Duration of postoperative drainage in subjects receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Duration of Postoperative Drainage in Gelfoam Plus Subjects: Duration of postoperative drainage in subjects receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Duration of Postoperative Drainage in BioFoam Subjects | Duration of Postoperative Drainage in Gelfoam Plus Subjects
Number analyzed (Participants) | 0 | 1
hours |  | NA — Study terminated before appropriate data collection/analysis

8. Secondary Outcome: Amount of Intraoperative Blood Products Administered
Description: Amount of blood products administered intraoperatively (throughout procedure: from initial skin cut to final wound closure)
Time Frame: Intraoperatively (throughout procedure, from initial skin cut to final wound closure, average 4-5 hours duration)
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: units of blood product(s)
Groups:
- Amt. of Intraop. Blood Products Rec'd by BioFoam Subjects: Amount of blood products administered intraoperatively to subjects receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Amt. of Intraop. Blood Products Rec'd by Gelfoam Plus Subjects: Amount of blood products administered intraoperatively to subjects receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Amt. of Intraop. Blood Products Rec'd by BioFoam Subjects | Amt. of Intraop. Blood Products Rec'd by Gelfoam Plus Subjects
Number analyzed (Participants) | 0 | 1
units of blood product(s) |  | NA — Study terminated before appropriate data collection/analysis

9. Secondary Outcome: Subject Laboratory Evaluations
Description: Number of laboratory evaluations outside of range from preoperative assessments through final 2 year follow-up
Time Frame: Preoperatively through final 2 year follow-up
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: Number of participants with labs in rang
Groups:
- Laboratory Evaluations for BioFoam Subjects Out of Range: Number of out of range lab evaluations for subjects receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Laboratory Evaluations for Gelfoam Plus Subjects Out of Range: Number of out of range lab evaluations for subjects receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Laboratory Evaluations for BioFoam Subjects Out of Range | Laboratory Evaluations for Gelfoam Plus Subjects Out of Range
Number analyzed (Participants) | 0 | 1
Number of participants with labs in rang |  | NA — Study terminated before appropriate data collection/analysis

10. Secondary Outcome: Eval. for Presence of Device by MRI w/ & w/Out Contrast, & Diagnose/Eval. Abdominal Fluid Collection/Biliary Leak, Residual Scarring, Hepatic Regeneration, & Assess for Emergence of Primary/Recurrent Malignancy by MRI w/ or w/Out Contrast as Appropriate
Time Frame: Within 48 hours postoperatively, up to 48 hours prior to hospital discharge (avg. 5-7 days postoperatively), and 30 days, 3 months, 6 months, 9 months, 1 year, and 2 years postoperatively
Measure: Number; unit: participants
Groups:
- Presence of Device Via MRI in BioFoam Surgical Matrix Subjects: Evaluation for presence of device via magnetic resonance imaging (MRI) in subjects receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Presence of Device Via MRI in Gelfoam Plus Subjects: Evaluation for presence of device via magnetic resonance imaging (MRI) in subjects receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Presence of Device Via MRI in BioFoam Surgical Matrix Subjects | Presence of Device Via MRI in Gelfoam Plus Subjects
Number analyzed (Participants) | 0 | 1
participants |  | 1

11. Secondary Outcome: Number of Subjects Requiring Reoperation Due to Bleeding and/or Biliary Leakage (Reoperation Required? y/n)
Description: Number of subjects requiring reoperation due to bleeding and/or biliary leakage out to 2 years postoperatively (reoperation required? y/n)
Time Frame: After final wound closure through 2 year follow-up visit (average 2 yr duration)
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: number of participants
Groups:
- BioFoam Subj. Requiring Reop. Due to Bleeding/Biliary Leakage: Number of subjects requiring reoperation due to bleeding and/or biliary leakage in subjects who received BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Gelfoam Plus Subj. Requiring Reop. Due to Bleeding/Bili. Leak: Number of subjects requiring reoperation due to bleeding and/or biliary leakage in subjects who received Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | BioFoam Subj. Requiring Reop. Due to Bleeding/Biliary Leakage | Gelfoam Plus Subj. Requiring Reop. Due to Bleeding/Bili. Leak
Number analyzed (Participants) | 0 | 1
number of participants |  | 0

12. Secondary Outcome: Total Time of Operative Procedure
Time Frame: Skin cut to skin closure (average 4-5 hour duration)
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: minutes
Groups:
- Total Time of Procedure for BioFoam Surgical Matrix Subjects: Total time of procedure for subjects receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Total Time of Procedure for Gelfoam Plus Subjects: Total time of procedure for subjects receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Total Time of Procedure for BioFoam Surgical Matrix Subjects | Total Time of Procedure for Gelfoam Plus Subjects
Number analyzed (Participants) | 0 | 1
minutes |  | 300

13. Secondary Outcome: Core Body Temperature
Time Frame: At the time of test or control article application (expected average 3-4 hours from skin cut)
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: degrees Celcius
Groups:
- Core Body Temp of BioFoam Subjects During Hemostat Application: Core body temp during prescribed topical hemostat application for subjects receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Core Body Temp of Gelfoam Plus During Hemostat Application: Core body temp during prescribed topical hemostat application for subjects receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Core Body Temp of BioFoam Subjects During Hemostat Application | Core Body Temp of Gelfoam Plus During Hemostat Application
Number analyzed (Participants) | 0 | 1
degrees Celcius |  | 36.5

14. Secondary Outcome: Total Hospitalization Time
Description: Length of time between hospital admission (day of surgery) and hospital discharge (average 5-7 days)
Time Frame: Hospital admission (day of surgery) until hospital discharge (average 5-7 days)
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: days
Groups:
- Length of Hospital Stay for BioFoam Surgical Matrix Subjects: Length of hospital stay for subjects receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Length of Hospital Stay for Gelfoam Plus Subjects: Length of hospital stay for subjects receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Length of Hospital Stay for BioFoam Surgical Matrix Subjects | Length of Hospital Stay for Gelfoam Plus Subjects
Number analyzed (Participants) | 0 | 1
days |  | NA — Study terminated before appropriate data collection/analysis

15. Secondary Outcome: Subjects Requiring Additional Hospitalization/Surgical Intervention
Description: Number of subjects requiring additional hospitalization/surgical intervention following final wound closure through the 2 year follow-up
Time Frame: Any hospitalization/surgical intervention following final wound closure through 2 year follow-up visit (average 2 yr duration)
Population: Study terminated before any subjects were enrolled into the BioFoam arm
Measure: Number; unit: # of participants
Groups:
- # of BioFoam Subjects Requiring Hospitalization/Intervention: Number of subjects receiving BioFoam Surgical Matrix as a surgical adjunct that required hospitalization or intervention following final wound closure through the 2 year follow-up visit
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- # of Gelfoam Plus Subj. Requiring Hospitalization/Intervention: Number of subjects receiving Gelfoam Plus as a surgical adjunct that required hospitalization or intervention following final wound closure through the 2 year follow-up visit
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | # of BioFoam Subjects Requiring Hospitalization/Intervention | # of Gelfoam Plus Subj. Requiring Hospitalization/Intervention
Number analyzed (Participants) | 0 | 1
# of participants |  | NA — Study terminated before appropriate data collection/analysis

16. Secondary Outcome: Evaluation of Anti-Bovine Serum Albumin (Anti-BSA) Antibody Titers
Description: Evaluation of anti-BSA antibody titers to determine number of subjects/participants with a positive titer at various time points
Time Frame: Preoperatively (up to 30 days before surgery), immediately post-application of hemostatic agent (within minutes), within 48 hrs postoperatively, up to 48 hrs before hospital discharge, at 7-10 days, 30 days, 3 mos, 6 mos, 9 mos, 1 yr, and 2 yr postop
Population: Blood samples were to be analyzed in batches to more accurately assess for any changes over time; the study was terminated before the first batch was analyzed, so no data is available for anti-BSA titer testing.
Groups:
- Anti-Bovine Serum Albumin (Anti-BSA) Titers in BioFoam Subj: Evaluation of anti-bovine serum albumin (anti-BSA) antibodies in subjects receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Anti-Bovine Serum Albumin (Anti-BSA) Titer in Gelfoam Plus Sub: Evaluation of anti-bovine serum albumin (anti-BSA) antibodies in subjects receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Anti-Bovine Serum Albumin (Anti-BSA) Titers in BioFoam Subj | Anti-Bovine Serum Albumin (Anti-BSA) Titer in Gelfoam Plus Sub
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Procedure Complications and/or Adverse Events
Time Frame: Through final follow-up (2 years postoperatively)
Measure: Number; unit: Number of complications and AEs
Groups:
- Complications/Adverse Events in Subjects Receiving BioFoam: Number of complications/adverse events recorded for subjects receiving BioFoam Surgical Matrix as a surgical adjunct
  BioFoam Surgical Matrix : Surgical adjunct to control bleeding in open liver surgery
- Complications/Adverse Events in Subj. Receiving Gelfoam Plus: Number of complications/adverse events recorded for subjects receiving Gelfoam Plus as a surgical adjunct
  Gelfoam Plus : Surgical adjunct in control of bleeding in open liver surgery
Arm/Group | Complications/Adverse Events in Subjects Receiving BioFoam | Complications/Adverse Events in Subj. Receiving Gelfoam Plus
Number analyzed (Participants) | 0 | 1
Number of complications and AEs |  | 31

ADVERSE EVENTS:
Arm/Group | BioFoam Surgical Matrix | Gelfoam Plus
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioFoam Surgical Matrix (N=0) | Gelfoam Plus (N=1)
Recurrence of Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Control subject, recurrence of hepatocellular carcinoma. Treatment of TACE with Cisplatin 12mg/Doxorubicin 12mg. Deemed as grade 2 (moderate) in severity, not related to either the study device or procedure. Event resolved with treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioFoam Surgical Matrix (N=0) | Gelfoam Plus (N=1)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abnormal Monocyte Count (Surgical and medical procedures) | 0 (0) | 1 (1)
Elevated AST (Surgical and medical procedures) | 0 (0) | 1 (1)
Elevated Total Protein (Surgical and medical procedures) | 0 (0) | 1 (1)
Hepatic Nodules (Hepatobiliary disorders) | 0 (0) | 1 (1)
High ALT (Surgical and medical procedures) | 0 (0) | 1 (1)
High Fibrinogen (Surgical and medical procedures) | 0 (0) | 1 (1)
High GGTP (Surgical and medical procedures) | 0 (0) | 1 (1)
High LDH (Surgical and medical procedures) | 0 (0) | 1 (1)
High WBC (Surgical and medical procedures) | 0 (0) | 1 (1)
Incisional Pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Intermittent Changes in Neutrophil Count (High) (Surgical and medical procedures) | 0 (0) | 1 (1)
Liver Function Tests Elevated ALT & AST (Surgical and medical procedures) | 0 (0) | 1 (1)
Low Bilirubin, Total (Surgical and medical procedures) | 0 (0) | 1 (1)
Low Calcium (Surgical and medical procedures) | 0 (0) | 1 (1)
Low Cholesterol (Surgical and medical procedures) | 0 (0) | 1 (1)
Low Creatinine (Surgical and medical procedures) | 0 (0) | 1 (1)
Low HGB (Surgical and medical procedures) | 0 (0) | 1 (1)
Low Lipase (Surgical and medical procedures) | 0 (0) | 1 (1)
Low Pancreatic Amylase (Surgical and medical procedures) | 0 (0) | 1 (1)
Low Phosphorus (Surgical and medical procedures) | 0 (0) | 1 (1)
Low Sodium (Surgical and medical procedures) | 0 (0) | 1 (1)
Low WBC (Surgical and medical procedures) | 0 (0) | 1 (1)
Lower Extremity Edema (General disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Worsened Baseline Low HCT (Surgical and medical procedures) | 0 (0) | 1 (1)
Worsened Baseline Low RBC (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects evaluated (n=1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship of 1st publication (Primary Paper) determined by Sponsor. If Primary Paper not sub. for publication within 18 months of study completion, Investigator may publish individual publication/presentation - proposal must be provided to Sponsor for review and comment at least 30 days prior to submission date/public disclosure. Sponsor to review within 30 days of receipt and can remove proprietary/confidential info and/or require delay in publication or public disclosure for up to 30 days.